CLINICAL TRIAL: NCT00332462
Title: A Multicenter, Open-label, Exploratory Study to Evaluate the Efficiency of Intravenously Administered Cyclosporine During the First 7 Days Post Transplant Followed by Treatment With Cyclosporine Micro Emulsion in de Novo Liver Transplant Recipients
Brief Title: A Study to Evaluate the Efficiency of Intravenously Administered Cyclosporine in de Novo Liver Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COLO400ADE01
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Results first posted 2011-01-11 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Liver Transplantation
Keywords: Liver transplantation, Cyclosporine
MeSH Terms: interventions — Cyclosporine

ARMS (1):
- Cyclosporine (Sandimmun®) (Experimental): Period 1: Cyclosporine (Sandimmun® i.v.) intravenous given 2 times daily as an infusion over four hours staring at a dose of 2 X 200 mg/day for 7 days followed by Period 2: Sandimmun® Optoral microemulsion oral capsule twice daily starting at an initial daily dose of 8-12 mg/kg/day. Dosages were adjusted based on blood levels at two hours to achieve protocol specified target levels.
  Interventions: Drug: Cyclosporine (Sandimmun® i.v.); Drug: Cyclosporine (Sandimmun® Optoral)

INTERVENTIONS:
Drug: Cyclosporine (Sandimmun® i.v.) — Cyclosporine (Sandimmun® i.v.) intravenous given 2 times daily as an infusion over four hours staring at a dose of 2 X 200 mg/day for 7 days. Dosages were adjusted based on blood levels at two hours to achieve protocol specified target levels.
  Other Names: Sandimmun
Drug: Cyclosporine (Sandimmun® Optoral) — Sandimmun® Optoral microemulsion oral capsule twice daily starting at an initial daily dose of 8-12 mg/kg/day. Dosages were adjusted based on blood levels at two hours to achieve protocol specified target levels.
  Other Names: Sandimmun

SUMMARY:
The aim of this exploratory study is to evaluate the rejection rate in patients treated with cyclosporine (CsA) preceding oral administration of cyclosporine micro emulsion in de novo liver recipients. The blood levels of CsA and CsA micro emulsion will be monitored by C-2h monitoring. In addition, this study will assess the safety of this treatment regimen.

ELIGIBILITY:
Inclusion Criteria

* About to undergo a primary liver transplant (including living donor, split liver).
* Expected to be capable of study participation for full 6 months post-transplantation.
* Allograft biopsies will be possible.

Exclusion Criteria

* The surgery is a multi-organ transplant.
* The patient has previously been transplanted with any other organ.
* The graft derives from a non-heart beating donor.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-05; Primary Completion 2008-04 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis Investigational Site, Various Cities, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cyclosporine (Sandimmun®)
Started | 34 (Safety and Intention to treat population.)
Patients Treated With Sandimmun® i.v. | 34
Patients Treated With Sandimmun® Optoral | 29
Completed | 18
Not Completed | 16
Not completed — Adverse Event | 5
Not completed — Abnormal Lab Value | 1
Not completed — Unsatisfactory therapeutic effect | 4
Not completed — no longer requires study drug | 1
Not completed — Death | 3
Not completed — Graft Loss | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cyclosporine (Sandimmun®)
Number analyzed (Participants) | 34
Age Continuous [Mean (Standard Deviation); unit: years] | 53.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Biopsy Proven Acute Rejection During the First 3 Months Post de Novo Liver Transplantation
Description: Number of patients with biopsy proven acute rejection (BPAR) within 3 months after post de novo liver transplantation. In all suspected rejection episodes an allograft biopsy was performed within a 48 hour period of initiation of an anti-rejection therapy. A designated pathologist graded the biopsies according to the Banff criteria into mild, moderate or severe BPAR.
Time Frame: 3 months
Population: Intention to treat (ITT) population
Measure: Number; unit: Participants
Arm/Group | Cyclosporine (Sandimmun®)
Number analyzed (Participants) | 34
Participants
  patients with BPAR within 3 months after Tx : YES | 8
  patients with BPAR within 3 months after Tx : NO | 26

2. Secondary Outcome: Incidence, Safety and Tolerability of Cyclosporine Intravenous (i.v.) During 6 Months Post de Novo Liver Transplantation
Description: The secondary efficacy endpoints included: the incidence of BPAR at 6 months; the incidence of treated acute rejection (TAR) / steroid-resistant acute rejection at 3 and 6 months; the incidence of BPAR with moderate/severe histological grading at 3 and 6 months; time to the first BPAR, the first TAR / steroid-resistant acute rejection and BPAR with moderate/severe histological grading; patient death at 3 and 6 months; and graft loss at 3 and 6 months.
Time Frame: 3 or 6 months after transplantation
Population: Intention-to-treat (ITT) population.
Measure: Number; unit: Participants
Arm/Group | 3 Months After Transplantation | 6 Months After Transplantation
Number analyzed (Participants) | 34 | 34
Participants
  Patients with BPAR : YES | NA — analysis was done for 6 month only | 10
  Patients with BPAR : NO | NA — analysis was done for 6 month only | 24
  Patients with TAR : YES | 7 | 8
  Patients with TAR : NO | 27 | 26
  Patients w/ steroid-resistant acute rejection:YES | 2 | 3
  Patients w/ steroid-resistant acute rejection:NO | 32 | 31
  BPAR w/ moderate/severe histological grading:YES | 4 | 4
  BPAR w/ moderate/severe histological grading:NO | 30 | 30
  Occurence of Death : YES | 3 | 3
  Occurence of Death : NO | 31 | 31
  Occurence of Graft loss : YES | 3 | 3
  Occurence of Graft loss : NO | 31 | 31

ADVERSE EVENTS:
Description: 34 of the 34 study participants received treatment with Cyclosporine (Sandimmun® i.v.). Only 29 of the 34 participants received treatment with Cyclosporine (Sandimmun® Optoral).
Groups:
- Cyclosporine (Sandimmun® i.v.): Cyclosporine (Sandimmun®) intravenous (i.v) given 2 times daily as an infusion over a four hour period staring at a dose of 2 X 200 mg/day and continuing for 7 days. Dosages were adjusted based on blood levels at two hours to achieve protocol specified target levels.
Arm/Group | Cyclosporine (Sandimmun® i.v.) | Cyclosporine (Sandimmun® Optoral)
Serious Adverse Events (participants affected / at risk) | 18/34 | 14/29
Other Adverse Events (participants affected / at risk) | 34/34 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine (Sandimmun® i.v.) (N=34) | Cyclosporine (Sandimmun® Optoral) (N=29)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0
ASCITES (Gastrointestinal disorders) | 0 | 2
PERITONEAL HAEMATOMA (Gastrointestinal disorders) | 1 | 0
HERNIA (General disorders) | 0 | 1
MULTI-ORGAN FAILURE (General disorders) | 1 | 0
SYSTEMIC LEAKAGE (General disorders) | 0 | 1
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 | 1
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 | 1
BILIARY ISCHAEMIA (Hepatobiliary disorders) | 0 | 2
CHOLANGITIS (Hepatobiliary disorders) | 0 | 3
CHOLANGITIS SCLEROSING (Hepatobiliary disorders) | 0 | 1
GRAFT VERSUS HOST DISEASE (Immune system disorders) | 0 | 1
LIVER TRANSPLANT REJECTION (Immune system disorders) | 0 | 1
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 0 | 1
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1 | 0
DIARRHOEA INFECTIOUS (Infections and infestations) | 0 | 1
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 1
HEPATITIS B (Infections and infestations) | 0 | 1
INFECTION (Infections and infestations) | 0 | 2
PNEUMONIA (Infections and infestations) | 1 | 1
SEPSIS (Infections and infestations) | 1 | 0
ABDOMINAL WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 1
COMPLICATIONS OF TRANSPLANTED LIVER (Injury, poisoning and procedural complications) | 2 | 1
HEPATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 | 1
SEROMA (Injury, poisoning and procedural complications) | 0 | 1
FIBRINOLYSIS INCREASED (Investigations) | 1 | 0
HEPATIC ENZYME INCREASED (Investigations) | 0 | 1
HEPATITIS C VIRUS (Investigations) | 0 | 1
NEUROENDOCRINE TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
ANURIA (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 2 | 2
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 | 1
HAEMORRHAGE (Vascular disorders) | 5 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine (Sandimmun® i.v.) (N=34) | Cyclosporine (Sandimmun® Optoral) (N=29)
ANAEMIA (Blood and lymphatic system disorders) | 18 | 10
COAGULOPATHY (Blood and lymphatic system disorders) | 12 | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 4
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 2
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 10 | 2
ARRHYTHMIA (Cardiac disorders) | 2 | 0
BRADYCARDIA (Cardiac disorders) | 5 | 1
TACHYARRHYTHMIA (Cardiac disorders) | 4 | 0
ANTITHROMBIN III DEFICIENCY (Congenital, familial and genetic disorders) | 8 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 8
ASCITES (Gastrointestinal disorders) | 2 | 4
CONSTIPATION (Gastrointestinal disorders) | 15 | 7
DIARRHOEA (Gastrointestinal disorders) | 2 | 7
FLATULENCE (Gastrointestinal disorders) | 4 | 3
NAUSEA (Gastrointestinal disorders) | 2 | 2
PERITONITIS (Gastrointestinal disorders) | 0 | 2
VOMITING (Gastrointestinal disorders) | 4 | 4
IMPAIRED HEALING (General disorders) | 0 | 5
MALAISE (General disorders) | 2 | 1
OEDEMA (General disorders) | 3 | 5
OEDEMA PERIPHERAL (General disorders) | 0 | 7
PUNCTURE SITE PAIN (General disorders) | 0 | 3
PYREXIA (General disorders) | 4 | 8
CHOLANGITIS (Hepatobiliary disorders) | 2 | 7
CHOLESTASIS (Hepatobiliary disorders) | 20 | 10
ABDOMINAL INFECTION (Infections and infestations) | 0 | 2
CANDIDIASIS (Infections and infestations) | 1 | 2
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1 | 5
FUNGAL INFECTION (Infections and infestations) | 0 | 2
HERPES SIMPLEX (Infections and infestations) | 1 | 2
INFECTION (Infections and infestations) | 5 | 2
PHARYNGITIS (Infections and infestations) | 1 | 2
PNEUMONIA (Infections and infestations) | 2 | 1
SEPSIS (Infections and infestations) | 3 | 0
SYSTEMIC CANDIDA (Infections and infestations) | 0 | 2
URINARY TRACT INFECTION (Infections and infestations) | 3 | 5
WOUND INFECTION (Infections and infestations) | 1 | 5
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 2 | 0
COMPLICATIONS OF TRANSPLANTED LIVER (Injury, poisoning and procedural complications) | 3 | 1
OPERATIVE HAEMORRHAGE (Injury, poisoning and procedural complications) | 5 | 0
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 3 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 17 | 2
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 2 | 4
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 | 2
TRANSAMINASES INCREASED (Investigations) | 1 | 3
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 2
FOLATE DEFICIENCY (Metabolism and nutrition disorders) | 0 | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 17 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 6 | 2
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 3
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 15 | 3
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 8 | 10
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 11 | 2
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 5
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 10 | 0
VITAMIN K DEFICIENCY (Metabolism and nutrition disorders) | 0 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 5
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 2
HEADACHE (Nervous system disorders) | 0 | 2
DEPRESSION (Psychiatric disorders) | 2 | 4
INSOMNIA (Psychiatric disorders) | 13 | 8
PSYCHOTIC DISORDER (Psychiatric disorders) | 4 | 0
SLEEP DISORDER (Psychiatric disorders) | 4 | 0
OLIGURIA (Renal and urinary disorders) | 5 | 0
RENAL FAILURE (Renal and urinary disorders) | 18 | 7
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 7 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 16 | 4
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 6 | 1
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 3 | 1
SCAR PAIN (Skin and subcutaneous tissue disorders) | 0 | 3
HAEMATOMA (Vascular disorders) | 2 | 0
HYPERTENSION (Vascular disorders) | 11 | 7
HYPOTENSION (Vascular disorders) | 17 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.